CLINICAL TRIAL: NCT02769923
Title: Intradermal Administration of Fractional Dose of Inactivated Poliovirus Vaccine Using Intradermal Adapters vs. BCG Syringe: Community Based Randomized Control Trial in Pakistan
Brief Title: ID Administration of fIPV Using Intradermal Adapters vs. BCG Syringe
Acronym: ID-ADAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, Ali Faisal Saleem, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3519-Ped-ERC-15
Record Dates: First submitted 2016-05-02; First posted 2016-05-12 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: IPV
Keywords: WestPharma ID-adapter; Star ID syringe; BCG needle syringe; fractional dose IPV; fIPV; polio; Polio Endgame; IPV
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (Active Comparator): Westpharma ID Adapter
  Interventions: Device: Westpharma ID adapter
- Arm B (Active Comparator): Star ID syringe
  Interventions: Device: Star ID syringe
- Arm C (Active Comparator): BCG NS
  Interventions: Device: BCG NS

INTERVENTIONS:
Device: Westpharma ID adapter — device used for administering intradermal injection
  Arms: Arm A
Device: Star ID syringe — device used for administering intradermal injection
  Arms: Arm B
Device: BCG NS — syringe used for administering intradermal injection
  Arms: Arm C

SUMMARY:
The investigators will assess the usability and immune response following fractional dose inactivated polio virus vaccine (fIPV) administration with two novel intradermal adapters (ID adapter by West Pharmaceutical services Inc. and Star Intradermal syringe by Star Syringe Ltd.) and compare the response with the one achieved with fIPV administered with traditional BCG needle syringe.

DETAILED DESCRIPTION:
The study will be conducted in following two phases.

1. Phase I: Ergonometric evaluation and serology: Phase I is based on community based randomized controlled trial with three arms. List of households with child aged 6-12 months will be retrieved from demographic surveillance system. Train CHWs will visit the household and provide relevant information regarding the study to the parents. The children of the parents who provide written informed consent will be screened for eligibility and enrolled into the study. The children accompanied with parents/guardians will be carried to the primary health center of the Dept. of pediatrics and child health, AKU. Baseline 3ml of blood will be collected by trained study phlebotomist in EDT tubes and will be transported to infectious disease research laboratory (IDRL) at AKU. A sample of 450 children will be randomized using sealed envelopes into one of the three study arms. Arm 1, will receive fIPV using WestPharma device, arm 2 will receive fIPV using Star ID syringe and arm 3 will receive fIPV using BCG syringe. The child will be observed for 30 minutes for any adverse event. The research Assistants will interview the parents to fill the socio-demographic questionnaire and vaccinators will fill ergonometric and injection quality questionnaires. The child will be followed after 28 days (4 weeks) of enrollment and another 3ml of blood will be collected by trained phlebotomist. Details of the visit will be recorded in follow-up questionnaire. Both baseline and endline blood samples will be tested for immune response against polio virus 1,2 and 3.
2. Phase II: Pilot campaign demonstration: In this phase, investigators will conduct a door to door campaign in the high risk community to provide fIPV using either WestPharma device or Star ID syringe or BCG needle syringe. In this campaign, any child less than 5 years of age, living in the study area and whose parents provide verbal consent will receive intradermal injection of fIPV using any of the three devices by the trained research assistants. This will be a one day campaign in coordination with provincial polio emergency operation center (EOC). About 300 children will receive fIPV using any of the three devices.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-12 months living in four peri-urban slums of Bin Qasim Town, Karachi (Rehri Goth, Bhains Colony, Ali Akber Shah, Ibrahim Hydri).

Exclusion Criteria:

* Child found acutely ill at the time of enrolment and requiring emergent medical care/hospitalization.
* Refusal of blood testing.
* Any contraindication for ID injection.
* A diagnosis or suspicion of immunodeficiency disorder (either in the participant or in a member of the immediate family.

  * e.g. several early infant deaths, household member on chemotherapy) will render the newborn ineligible for the study.

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 450 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Difference in immune response against poliovirus type 1, 2 and 3 after 28 days of administration of fractional dose IPV | up to day 28.
  Seropositivity is defined as reciprocal titers of poliovirus neutralizing antibodies >8; seroconversion is defined as the change from seronegative to seropositive (from reciprocal titer of <8 to >8); and boosting is defined as >4-fold increase in titers. In this study, "immune response" combines both boosting and seroconversion.

SECONDARY OUTCOMES:
Difference in bleb size after the intradermal injection among three arms | immediately after injection
  The bleb size will measured immediately after the administration of injection using the millimeter scale.
Difference in vaccine loss after the intradermal injection among three arms | immediately after injection
  The measurement is performed by blotting the skin with filter paper to collect liquid that was not delivered into the skin or leaked out after injection. The wet spot on the filter paper will be circled and the diameter of the circle compared to a reference template to quantify the amount of liquid present into the following categories: 0 μl, 0 to 5 μl, 5 to 10 μl, 10 to 20 μl, 20 to 40 μl, more than 40 μl.
Difference in local adverse events | within 30 minutes after injection
  local adverse events include redness, itching, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Ali F Saleem, FCPS,MSc, Principal Investigator — The Aga Khan University, Karachi; Mohammad T Yousafzai, MPH, MSc, Principal Investigator — The Aga Khan University, Karachi

IPD SHARING:
Plan to Share IPD: Yes
in process